CLINICAL TRIAL: NCT02285504
Title: An Open-Label Proof-of-Concept Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of SAGE-547 Injection in the Treatment of Adult Female Patients With Severe Postpartum Depression
Brief Title: Evaluate SAGE-547 in Female Participants With Severe Postpartum Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 547-PPD-201
Record Dates: First submitted 2014-10-22; First posted 2014-11-07 (Estimated); Results first posted 2021-12-02 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2021-11

CONDITIONS: Postpartum Depression
Keywords: Postpartum depression
MeSH Terms: conditions — Depression, Postpartum | interventions — brexanolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SAGE-547 (Experimental): Participants received SAGE-547 intravenous injection over 60 hours (including 12-hour titration infusion of 21.5 micrograms per kilogram per hour [mcg/kg/hr] [4 hrs], 43 mcg/kg/hr [4 hrs] and 64.5 mcg/kg/hr [4 hrs] on Day 1, followed by 13 to 48 hrs [36 hrs] maintenance infusion of 86 mcg/kg/hr from Day 1 to 3, followed by a 12-hr taper infusion of 64.5 mcg/kg/hr [49 - 52 hrs], 43 mcg/kg/hr [53 - 56 hrs] and 21.5 mcg/kg/hr [57 - 60 hrs] on Day 3).
  Interventions: Drug: SAGE-547

INTERVENTIONS:
Drug: SAGE-547 — Intravenous injection

SUMMARY:
This is an open-label proof-of-concept study designed to evaluate the safety, tolerability, pharmacokinetics (PK), and efficacy of SAGE-547 Injection in adult female participants diagnosed with severe postpartum depression (PPD).

ELIGIBILITY:
Inclusion Criteria:

* Adult females, 18-45 years old who experienced a major depressive episode in the postpartum period beginning within the first 4 weeks following delivery
* Participant has ceased lactating, or if still lactating has already fully and permanently weaned their infant; if still actively breastfeeding, participant must agree to cease giving breast milk to their infant prior to study entry

Exclusion Criteria:

* Recent history or active clinically significant manifestations of metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, musculoskeletal, dermatological, urogenital, or eyes, ears, or nose and throat (EENT) disorders
* Active psychosis
* Medical history of seizures

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2015-01-07 (Actual); Primary Completion 2015-06-05 (Actual); Study Completion 2015-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Kanes, MD, PhD, Study Chair — Sage Therapeutics
Locations (1):
- Sage Investigational Site, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.

REFERENCES:
- See also: Sage Therapeutics — http://www.sagerx.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study at 1 center in the United States from 07 January 2015 to 05 June 2015.
Pre-assignment Details: A total of 6 participants were screened, 4 participants were treated and completed the study. This study consisted of up to a 3-day screening period, a 4-day (84-hour) active treatment period, a 7-day adverse event (AE) follow-up period, plus an additional 23 days of serious AE follow-up (with a telephone call at Day 11 and Day 34).
Period: Overall Study
Arm/Group | SAGE-547
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who began infusion with SAGE-547 injection.
Groups:
- SAGE-547: Participants received SAGE-547 intravenous injection over 60 hours (including 12-hour titration infusion of 21.5 mcg/kg/hr [4 hrs], 43 mcg/kg/hr [4 hrs] and 64.5 mcg/kg/hr [4 hrs] on Day 1, followed by 13 to 48 hrs [36 hrs] maintenance infusion of 86 mcg/kg/hr from Day 1 to 3, followed by a 12-hr taper infusion of 64.5 mcg/kg/hr [49 - 52 hrs], 43 mcg/kg/hr [53 - 56 hrs] and 21.5 mcg/kg/hr [57 - 60 hrs] on Day 3).
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.0 (6.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: AEs were any untoward medical occurrences in a participant who received study treatment without regard to possibility of causal relationship. TEAEs were defined as AEs with onset after the start of SAGE-547 infusion, or any worsening of a pre-existing medical condition or AEs with onset after the start of SAGE-547 infusion and until 7 days after the end of infusion (Day 11). TESAEs were defined as AEs with onset after the start of SAGE-547 infusion, or any worsening of a pre-existing medical condition or AEs with onset after the start of SAGE-547 infusion and until 30 days after the end of infusion (Day 34).
Time Frame: TEAEs: Up to Day 11, TESAEs: Up to Day 34
Population: Safety population included all participants who began infusion with SAGE-547 injection.
Measure: Count of Participants; unit: Participants
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
Participants
  TEAEs | 4
  TESAEs | 0

2. Primary Outcome: Change From Baseline in Clinical Laboratory Measures: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Gamma Glutamyl Transferase (GGT)
Description: Clinical laboratory evaluation included: Chemistry (ALT, AST, GGT) expressed in terms of units per liter (U/L). The data was collected at time-points on Days 2 (at 24 hrs), 3 (at 48 hrs) and 4 (at 84 hrs).
Time Frame: Baseline, Days 2 (at 24 hrs), 3 (at 48 hrs) and 4 (at 84 hrs)
Population: Safety population included all participants who began infusion with SAGE-547 injection. Here, 'number analyzed' signifies participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
U/L
  Change From Baseline at Day 2 (24 hrs): ALT | -3.0 (4.69)
  Change From Baseline at Day 3 (48 hrs): ALT: number analyzed (Participants) | 3
  Change From Baseline at Day 3 (48 hrs): ALT | -3.7 (7.02)
  Change From Baseline at Day 4 (84 hrs): ALT: number analyzed (Participants) | 3
  Change From Baseline at Day 4 (84 hrs): ALT | 2.7 (2.08)
  Change From Baseline at Day 2 (24 hrs): AST | -0.5 (6.19)
  Change From Baseline at Day 3 (48 hrs): AST: number analyzed (Participants) | 3
  Change From Baseline at Day 3 (48 hrs): AST | 1.0 (6.24)
  Change From Baseline at Day 4 (84 hrs): AST: number analyzed (Participants) | 3
  Change From Baseline at Day 4 (84 hrs): AST | 4.7 (5.69)
  Change From Baseline at Day 2 (24 hrs): GGT: number analyzed (Participants) | 3
  Change From Baseline at Day 2 (24 hrs): GGT | -0.7 (2.08)
  Change From Baseline at Day 3 (48 hrs): GGT: number analyzed (Participants) | 2
  Change From Baseline at Day 3 (48 hrs): GGT | -2.0 (1.41)
  Change From Baseline at Day 4 (84 hrs): GGT: number analyzed (Participants) | 2
  Change From Baseline at Day 4 (84 hrs): GGT | 5.5 (9.19)

3. Primary Outcome: Change From Baseline in Clinical Laboratory Measures: Carbon Dioxide (CO2), Sodium, Potassium and Chloride
Description: Clinical laboratory evaluation included: Chemistry (carbon dioxide [CO2], sodium, potassium and chloride) expressed in terms of millimoles/liter (mmol/L). The data was collected at time-points on Days 2 (at 24 hrs), 3 (at 48 hrs) and 4 (at 84 hrs).
Time Frame: Baseline, Days 2 (at 24 hrs), 3 (at 48 hrs) and 4 (at 84 hrs)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
mmol/L
  Change From Baseline at Day 2 (24 hrs): CO2 | -0.5 (3.42)
  Change From Baseline at Day 3 (48 hrs): CO2: number analyzed (Participants) | 3
  Change From Baseline at Day 3 (48 hrs): CO2 | -2.0 (3.61)
  Change From Baseline at Day 4 (84 hrs): CO2: number analyzed (Participants) | 3
  Change From Baseline at Day 4 (84 hrs): CO2 | -3.0 (4.58)
  Change From Baseline at Day 2 (24 hrs): Sodium | -0.5 (1.00)
  Change From Baseline at Day 3 (48 hrs): Sodium: number analyzed (Participants) | 3
  Change From Baseline at Day 3 (48 hrs): Sodium | -1.3 (2.08)
  Change From Baseline at Day 4 (84 hrs): Sodium: number analyzed (Participants) | 3
  Change From Baseline at Day 4 (84 hrs): Sodium | 1.3 (2.52)
  Change From Baseline at Day 2 (24 hrs): Potassium | 0.25 (0.208)
  Change From Baseline at Day 3 (48 hrs): Potassium: number analyzed (Participants) | 3
  Change From Baseline at Day 3 (48 hrs): Potassium | 0.20 (0.100)
  Change From Baseline at Day 4 (84 hrs): Potassium: number analyzed (Participants) | 3
  Change From Baseline at Day 4 (84 hrs): Potassium | 0.47 (0.115)
  Change From Baseline at Day 2 (24 hrs): Chloride | -0.5 (5.00)
  Change From Baseline at Day 3 (48 hrs): Chloride: number analyzed (Participants) | 3
  Change From Baseline at Day 3 (48 hrs): Chloride | -1.3 (5.03)
  Change From Baseline at Day 4 (84 hrs): Chloride: number analyzed (Participants) | 3
  Change From Baseline at Day 4 (84 hrs): Chloride | -1.3 (6.03)

4. Primary Outcome: Change From Baseline in Clinical Laboratory Measures: Glucose, Total Bilirubin, Calcium, Blood Urea Nitrogen (BUN) and Creatinine
Description: Clinical laboratory evaluation included: Chemistry (glucose, total bilirubin, calcium, blood urea nitrogen [BUN] and creatinine) expressed in terms of milligrams/deciliter (mg/dL). The data was collected at time-points on Days 2 (at 24 hrs), 3 (at 48 hrs) and 4 (at 84 hrs).
Time Frame: Baseline, Days 2 (at 24 hrs), 3 (at 48 hrs) and 4 (at 84 hrs)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
mg/dL
  Change at Day 2 (24 hrs): Glucose | 16.0 (15.90)
  Change at Day 3 (48 hrs): Glucose: number analyzed (Participants) | 3
  Change at Day 3 (48 hrs): Glucose | 28.3 (31.37)
  Change at Day 4 (84 hrs): Glucose: number analyzed (Participants) | 3
  Change at Day 4 (84 hrs): Glucose | 17.7 (13.58)
  Change at Day 2 (24 hrs): Total Bilirubin | -0.05 (0.129)
  Change at Day 3 (48 hrs): Total Bilirubin: number analyzed (Participants) | 3
  Change at Day 3 (48 hrs): Total Bilirubin | -0.23 (0.153)
  Change at Day 4 (84 hrs): Total Bilirubin: number analyzed (Participants) | 3
  Change at Day 4 (84 hrs): Total Bilirubin | -0.13 (0.115)
  Change at Day 2 (24 hrs): Calcium | -0.28 (0.532)
  Change at Day 3 (48 hrs): Calcium: number analyzed (Participants) | 3
  Change at Day 3 (48 hrs): Calcium | -0.03 (0.802)
  Change at Day 4 (84 hrs): Calcium: number analyzed (Participants) | 3
  Change at Day 4 (84 hrs): Calcium | 0.30 (0.265)
  Change at Day 2 (24 hrs): BUN | 0.5 (1.29)
  Change at Day 3 (48 hrs): BUN: number analyzed (Participants) | 3
  Change at Day 3 (48 hrs): BUN | 0.3 (4.51)
  Change at Day 4 (84 hrs): BUN: number analyzed (Participants) | 3
  Change at Day 4 (84 hrs): BUN | 0.0 (4.58)
  Change at Day 2 (24 hrs): Creatinine | -0.010 (0.0698)
  Change at Day 3 (48 hrs): Creatinine: number analyzed (Participants) | 3
  Change at Day 3 (48 hrs): Creatinine | -0.050 (0.0721)
  Change at Day 4 (84 hrs): Creatinine: number analyzed (Participants) | 3
  Change at Day 4 (84 hrs): Creatinine | -0.057 (0.1159)

5. Primary Outcome: Change From Baseline in Clinical Laboratory Measures: Albumin, Total Protein and Hemoglobin
Description: Clinical laboratory evaluation included: Chemistry (albumin, total protein), Hematology and Coagulation (hemoglobin) expressed in terms of g/dL. The data was collected at time-points on Days 2 (at 24 hrs), 3 (at 48 hrs) and 4 (at 84 hrs).
Time Frame: Baseline, Days 2 (at 24 hrs), 3 (at 48 hrs) and 4 (at 84 hrs)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
g/dL
  Change at Day 2 (24 hrs): Albumin | -0.40 (0.497)
  Change at Day 3 (48 hrs): Albumin: number analyzed (Participants) | 3
  Change at Day 3 (48 hrs): Albumin | -0.33 (0.551)
  Change at Day 4 (84 hrs): Albumin: number analyzed (Participants) | 3
  Change at Day 4 (84 hrs): Albumin | 0.20 (0.173)
  Change at Day 2 (24 hrs): Total Protein | -0.63 (0.499)
  Change at Day 3 (48 hrs): Total Protein: number analyzed (Participants) | 3
  Change at Day 3 (48 hrs): Total Protein | -0.43 (0.702)
  Change at Day 4 (84 hrs): Total Protein: number analyzed (Participants) | 3
  Change at Day 4 (84 hrs): Total Protein | 0.20 (0.361)
  Change at Day 2 (24 hrs): Hemoglobin | 0.02 (0.943)
  Change at Day 3 (48 hrs): Hemoglobin: number analyzed (Participants) | 3
  Change at Day 3 (48 hrs): Hemoglobin | -0.10 (0.954)
  Change at Day 4 (84 hrs): Hemoglobin: number analyzed (Participants) | 3
  Change at Day 4 (84 hrs): Hemoglobin | 0.27 (0.306)

6. Primary Outcome: Change From Baseline in Clinical Laboratory Measure: Hematocrit
Description: Clinical laboratory evaluation included: Hematocrit expressed in terms of percentage. The data was collected at time-points on Days 2 (at 24 hrs), 3 (at 48 hrs) and 4 (at 84 hrs).
Time Frame: Baseline, Days 2 (at 24 hrs), 3 (at 48 hrs) and 4 (at 84 hrs)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of hematocrit
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
percentage of hematocrit
  Change From Baseline at Day 2 (24 hrs) | 0.15 (2.199)
  Change From Baseline at Day 3 (48 hrs): number analyzed (Participants) | 3
  Change From Baseline at Day 3 (48 hrs) | -1.07 (1.914)
  Change From Baseline at Day 4 (84 hrs): number analyzed (Participants) | 3
  Change From Baseline at Day 4 (84 hrs) | 1.20 (1.311)

7. Primary Outcome: Change From Baseline in Clinical Laboratory Measures: Platelet Count, White Blood Cells (WBC), Absolute Lymphocytes, Absolute Neutrophils, Absolute Basophils, Absolute Eosinophils, Absolute Monocytes
Description: Clinical laboratory evaluation included: Platelet count, white blood cells (WBC), absolute lymphocytes, absolute neutrophils, absolute basophils, absolute eosinophils, absolute monocytes expressed in terms of 10^9 cells/L. The data was collected at time-points on Days 2 (at 24 hrs), 3 (at 48 hrs) and 4 (at 84 hrs).
Time Frame: Baseline, Days 2 (at 24 hrs), 3 (at 48 hrs) and 4 (at 84 hrs)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
10^9 cells/L
  Change at Day 2 (24 hrs): Platelet Count | -18.8 (16.50)
  Change at Day 3 (48 hrs): Platelet Count: number analyzed (Participants) | 3
  Change at Day 3 (48 hrs): Platelet Count | -23.3 (27.65)
  Change at Day 4 (84 hrs): Platelet Count: number analyzed (Participants) | 3
  Change at Day 4 (84 hrs): Platelet Count | -4.3 (37.98)
  Change at Day 2 (24 hrs): WBC | -0.93 (1.910)
  Change at Day 3 (48 hrs): WBC: number analyzed (Participants) | 3
  Change at Day 3 (48 hrs): WBC | -0.03 (3.287)
  Change at Day 4 (84 hrs): WBC: number analyzed (Participants) | 3
  Change at Day 4 (84 hrs): WBC | -1.07 (1.069)
  Change at Day 2 (24 hrs): Absolute Lymphocytes: number analyzed (Participants) | 3
  Change at Day 2 (24 hrs): Absolute Lymphocytes | -0.73 (0.764)
  Change at Day 3 (48 hrs): Absolute Lymphocytes: number analyzed (Participants) | 2
  Change at Day 3 (48 hrs): Absolute Lymphocytes | -0.50 (1.273)
  Change at Day 4 (84 hrs): Absolute Lymphocytes: number analyzed (Participants) | 3
  Change at Day 4 (84 hrs): Absolute Lymphocytes | -0.57 (0.737)
  Change at Day 2 (24 hrs): Absolute Neutrophils: number analyzed (Participants) | 3
  Change at Day 2 (24 hrs): Absolute Neutrophils | -0.933 (0.2082)
  Change at Day 3 (48 hrs): Absolute Neutrophils: number analyzed (Participants) | 2
  Change at Day 3 (48 hrs): Absolute Neutrophils | -1.250 (0.2121)
  Change at Day 4 (84 hrs): Absolute Neutrophils: number analyzed (Participants) | 3
  Change at Day 4 (84 hrs): Absolute Neutrophils | -0.467 (0.2082)
  Change at Day 2 (24 hrs): Absolute Basophils: number analyzed (Participants) | 3
  Change at Day 2 (24 hrs): Absolute Basophils | 0.0 (0.00)
  Change at Day 3 (48 hrs): Absolute Basophils: number analyzed (Participants) | 2
  Change at Day 3 (48 hrs): Absolute Basophils | 0.0 (0.00)
  Change at Day 4 (84 hrs): Absolute Basophils: number analyzed (Participants) | 3
  Change at Day 4 (84 hrs): Absolute Basophils | 0.0 (0.00)
  Change at Day 2 (24 hrs): Absolute Eosinophils: number analyzed (Participants) | 3
  Change at Day 2 (24 hrs): Absolute Eosinophils | 0.03 (0.058)
  Change at Day 3 (48 hrs): Absolute Eosinophils: number analyzed (Participants) | 2
  Change at Day 3 (48 hrs): Absolute Eosinophils | 0.05 (0.071)
  Change at Day 4 (84 hrs): Absolute Eosinophils: number analyzed (Participants) | 3
  Change at Day 4 (84 hrs): Absolute Eosinophils | 0.00 (0.100)
  Change at Day 2 (24 hrs): Absolute Monocytes: number analyzed (Participants) | 3
  Change at Day 2 (24 hrs): Absolute Monocytes | -0.10 (0.100)
  Change at Day 3 (48 hrs): Absolute Monocytes: number analyzed (Participants) | 2
  Change at Day 3 (48 hrs): Absolute Monocytes | -0.05 (0.071)
  Change at Day 4 (84 hrs): Absolute Monocytes: number analyzed (Participants) | 3
  Change at Day 4 (84 hrs): Absolute Monocytes | -0.07 (0.058)

8. Primary Outcome: Change From Baseline in Clinical Laboratory Measure: Red Blood Cells (RBC)
Description: Clinical laboratory evaluation included: RBC expressed in terms of 10^12 cells/L. The data was collected at time-points on Days 2 (at 24 hrs), 3 (at 48 hrs) and 4 (at 84 hrs).
Time Frame: Baseline, Days 2 (at 24 hrs), 3 (at 48 hrs) and 4 (at 84 hrs)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
10^12 cells/L
  Change From Baseline at Day 2 (24 hrs) | -0.030 (0.1924)
  Change From Baseline at Day 3 (48 hrs): number analyzed (Participants) | 3
  Change From Baseline at Day 3 (48 hrs) | -0.090 (0.2784)
  Change From Baseline at Day 4 (84 hrs): number analyzed (Participants) | 3
  Change From Baseline at Day 4 (84 hrs) | 0.113 (0.1656)

9. Primary Outcome: Change From Baseline in Clinical Laboratory Measure: Mean Corpuscular Volume (MCV)
Description: Clinical laboratory evaluation included: MCV expressed in terms of femtoliters (fL). The data was collected at time-points on Days 2 (at 24 hrs), 3 (at 48 hrs) and 4 (at 84 hrs).
Time Frame: Baseline, Days 2 (at 24 hrs), 3 (at 48 hrs) and 4 (at 84 hrs)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
fL
  Change From Baseline at Day 2 (24 hrs) | 0.85 (1.578)
  Change From Baseline at Day 3 (48 hrs): number analyzed (Participants) | 3
  Change From Baseline at Day 3 (48 hrs) | -0.53 (0.924)
  Change From Baseline at Day 4 (84 hrs): number analyzed (Participants) | 3
  Change From Baseline at Day 4 (84 hrs) | 0.33 (1.155)

10. Primary Outcome: Change From Baseline in Clinical Laboratory Measure: Mean Corpuscular Hemoglobin (MCH)
Description: Clinical laboratory evaluation included: MCH expressed in terms of picogram (pg). The data was collected at time-points on Days 2 (at 24 hrs), 3 (at 48 hrs) and 4 (at 84 hrs).
Time Frame: Baseline, Days 2 (at 24 hrs), 3 (at 48 hrs) and 4 (at 84 hrs)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
pg
  Change From Baseline at Day 2 (24 hrs): number analyzed (Participants) | 3
  Change From Baseline at Day 2 (24 hrs) | -0.3 (1.15)
  Change From Baseline at Day 3 (48 hrs): number analyzed (Participants) | 2
  Change From Baseline at Day 3 (48 hrs) | 0.5 (0.71)
  Change From Baseline at Day 4 (84 hrs): number analyzed (Participants) | 3
  Change From Baseline at Day 4 (84 hrs) | -0.3 (1.15)

11. Primary Outcome: Change From Baseline in Clinical Laboratory Measure: Prothrombin Time/International Normalized Ratio (PT/INR)
Description: Clinical laboratory evaluation included: PT/INR expressed in terms of seconds. The data was collected at time-points on Days 2 (at 24 hrs), 3 (at 48 hrs) and 4 (at 84 hrs).
Time Frame: Baseline, Days 2 (at 24 hrs), 3 (at 48 hrs) and 4 (at 84 hrs)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
seconds
  Change From Baseline at Day 2 (24 hrs): number analyzed (Participants) | 3
  Change From Baseline at Day 2 (24 hrs) | -0.30 (0.700)
  Change From Baseline at Day 3 (48 hrs): number analyzed (Participants) | 2
  Change From Baseline at Day 3 (48 hrs) | -1.05 (0.636)
  Change From Baseline at Day 4 (84 hrs): number analyzed (Participants) | 3
  Change From Baseline at Day 4 (84 hrs) | -0.37 (0.902)

12. Primary Outcome: Change From Baseline in Clinical Laboratory Measure: Potential of Hydrogen (pH)
Description: Clinical laboratory evaluation included: Urinalysis (pH). The data was collected at time-points on Days 2 (at 24 hrs), 3 (at 48 hrs) and 4 (at 84 hrs).
Time Frame: Baseline, Days 2 (at 24 hrs), 3 (at 48 hrs) and 4 (at 84 hrs)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
pH
  Change From Baseline at Day 2 (24 hrs): number analyzed (Participants) | 3
  Change From Baseline at Day 2 (24 hrs) | -0.17 (1.155)
  Change From Baseline at Day 3 (48 hrs): number analyzed (Participants) | 3
  Change From Baseline at Day 3 (48 hrs) | 0.33 (0.289)
  Change From Baseline at Day 4 (84 hrs): number analyzed (Participants) | 2
  Change From Baseline at Day 4 (84 hrs) | 1.00 (0.000)

13. Primary Outcome: Change From Baseline in Clinical Laboratory Measure: Specific Gravity
Description: Clinical laboratory evaluation included: Urinalysis (specific gravity) expressed in terms of ratio. The data was collected at time-points on Days 2 (at 24 hrs), 3 (at 48 hrs) and 4 (at 84 hrs).
Time Frame: Baseline, Days 2 (at 24 hrs), 3 (at 48 hrs) and 4 (at 84 hrs)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
ratio
  Change From Baseline at Day 2 (24 hrs): number analyzed (Participants) | 3
  Change From Baseline at Day 2 (24 hrs) | -0.0080 (0.00458)
  Change From Baseline at Day 3 (48 hrs): number analyzed (Participants) | 3
  Change From Baseline at Day 3 (48 hrs) | -0.0017 (0.00252)
  Change From Baseline at Day 4 (84 hrs): number analyzed (Participants) | 2
  Change From Baseline at Day 4 (84 hrs) | -0.0015 (0.00495)

14. Primary Outcome: Change From Baseline in Vital Sign: Blood Pressure
Description: Vital sign parameters included supine systolic blood pressure (SBP), supine diastolic blood pressure (DBP), standing systolic blood pressure and standing diastolic blood pressure expressed in terms of millimeters of mercury (mmHg). The data was collected at time-points on Day 1 (12 hrs), Day 2 (at 24 and 36 hrs), on Day 3 (at 48 and 60 hrs), and Day 4 (at 72 and 84 hrs).
Time Frame: Baseline, Day 1 (12 hrs), Day 2 (at 24 and 36 hrs), on Day 3 (at 48 and 60 hrs), and Day 4 (at 72 and 84 hrs)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
mmHg
  Change From Baseline at Day 1 (12 hrs): Supine SBP | -2.8 (13.65)
  Change From Baseline at Day 2 (24 hrs): Supine SBP | 2.3 (11.95)
  Change From Baseline at Day 2 (36 hrs): Supine SBP | -1.0 (15.19)
  Change From Baseline at Day 3 (48 hrs): Supine SBP | -5.0 (4.40)
  Change From Baseline at Day 3 (60 hrs): Supine SBP | 12.3 (17.75)
  Change From Baseline at Day 4 (72 hrs): Supine SBP | 5.0 (23.73)
  Change From Baseline at Day 4 (84 hrs): Supine SBP | 8.0 (20.69)
  Change From Baseline at Day 1 (12 hrs): Supine DBP | -1.3 (12.50)
  Change From Baseline at Day 2 (24 hrs): Supine DBP | 3.0 (6.83)
  Change From Baseline at Day 2 (36 hrs): Supine DBP | -2.3 (5.68)
  Change From Baseline at Day 3 (48 hrs): Supine DBP | -5.0 (5.42)
  Change From Baseline at Day 3 (60 hrs): Supine DBP | 4.0 (6.22)
  Change From Baseline at Day 4 (72 hrs): Supine DBP | 0.5 (9.75)
  Change From Baseline at Day 4 (84 hrs): Supine DBP | 7.5 (10.21)
  Change From Baseline at Day 1(12 hrs):Standing SBP | -4.0 (7.87)
  Change From Baseline at Day 2(24 hrs):Standing SBP | -1.5 (8.23)
  Change From Baseline at Day 2(36 hrs):Standing SBP | -0.8 (7.27)
  Change From Baseline at Day 3(48 hrs):Standing SBP | -1.5 (7.68)
  Change From Baseline at Day 3(60 hrs):Standing SBP | 16.8 (2.50)
  Change From Baseline at Day 4(72 hrs):Standing SBP | 0.3 (11.53)
  Change From Baseline at Day 4(84 hrs):Standing SBP: number analyzed (Participants) | 3
  Change From Baseline at Day 4(84 hrs):Standing SBP | -0.7 (8.74)
  Change From Baseline at Day 1(12 hrs):Standing DBP | 1.0 (8.52)
  Change From Baseline at Day 2(24 hrs):Standing DBP | 6.3 (4.11)
  Change From Baseline at Day 2(36 hrs):Standing DBP | 1.5 (9.11)
  Change From Baseline at Day 3(48 hrs):Standing DBP | 7.5 (5.92)
  Change From Baseline at Day 3(60 hrs):Standing DBP | 13.8 (8.81)
  Change From Baseline at Day 4(72 hrs):Standing DBP | 13.3 (8.14)
  Change From Baseline at Day 4(84 hrs):Standing DBP: number analyzed (Participants) | 3
  Change From Baseline at Day 4(84 hrs):Standing DBP | 10.3 (3.06)

15. Primary Outcome: Change From Baseline in Vital Sign: Heart Rate
Description: Vital sign parameter included heart rate expressed in terms of beats per minute (bpm). The data was collected at time-points on Day 1 (12 hrs), Day 2 (at 24 and 36 hrs), on Day 3 (at 48 and 60 hrs), and Day 4 (at 72 and 84 hrs).
Time Frame: Baseline, Day 1 (12 hrs) Day 2 (at 24 and 36 hrs), on Day 3 (at 48 and 60 hrs), and Day 4 (at 72 and 84 hrs)
Population: Safety population included all participants who began infusion with SAGE-547 injection.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
bpm
  Change From Baseline at Day 1 (12 hrs) | -2.5 (15.35)
  Change From Baseline at Day 2 (24 hrs) | 5.3 (18.84)
  Change From Baseline at Day 2 (36 hrs) | -2.3 (11.44)
  Change From Baseline at Day 3 (48 hrs) | -1.5 (11.56)
  Change From Baseline at Day 3 (60 hrs) | -3.0 (8.41)
  Change From Baseline at Day 4 (72 hrs) | -5.8 (7.63)
  Change From Baseline at Day 4 (84 hrs) | -0.8 (4.99)

16. Primary Outcome: Change From Baseline in Vital Sign: Body Temperature
Description: Vital sign parameter included temperature expressed in terms of degree Celsius. The data was collected at time-points on Day 1 (12 hrs), Day 2 (at 24 and 36 hrs), on Day 3 (at 48 and 60 hrs), and Day 4 (at 72 and 84 hrs).
Time Frame: Baseline, Day 1 (12 hrs) Day 2 (at 24 and 36 hrs), on Day 3 (at 48 and 60 hrs), and Day 4 (at 72 and 84 hrs)
Population: Safety population included all participants who began infusion with SAGE-547 injection.
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
degree Celsius
  Change From Baseline at Day 1 (12 hrs) | -0.20 (0.32)
  Change From Baseline at Day 2 (24 hrs) | 0.15 (0.23)
  Change From Baseline at Day 2 (36 hrs) | -0.15 (0.33)
  Change From Baseline at Day 3 (48 hrs) | -0.05 (0.25)
  Change From Baseline at Day 3 (60 hrs) | 0.03 (0.31)
  Change From Baseline at Day 4 (72 hrs) | -0.30 (0.37)
  Change From Baseline at Day 4 (84 hrs) | -0.45 (0.46)

17. Primary Outcome: Change From Baseline in Vital Sign: Respiratory Rate
Description: Vital sign parameter included respiratory rate expressed in terms of breaths per minute. The data was collected at time-points on Day 1 (12 hrs), Day 2 (at 24 and 36 hrs), on Day 3 (at 48 and 60 hrs), and Day 4 (at 72 and 84 hrs).
Time Frame: Baseline, Day 1 (12 hrs) Day 2 (at 24 and 36 hrs), on Day 3 (at 48 and 60 hrs), and Day 4 (at 72 and 84 hrs)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
breaths/min
  Change From Baseline at Day 1 (12 hrs) | 0.0 (1.63)
  Change From Baseline at Day 2 (24 hrs) | 0.0 (2.31)
  Change From Baseline at Day 2 (36 hrs) | 0.0 (2.31)
  Change From Baseline at Day 3 (48 hrs) | 0.0 (4.00)
  Change From Baseline at Day 3 (60 hrs): number analyzed (Participants) | 3
  Change From Baseline at Day 3 (60 hrs) | 0.3 (1.53)
  Change From Baseline at Day 4 (72 hrs) | -1.0 (1.15)
  Change From Baseline at Day 4 (84 hrs) | -0.5 (1.00)

18. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters: QT Interval, PR Interval, QTc Interval, and QRS Duration
Description: ECGs parameters included QT interval, PR interval, QTc interval, QRS duration expressed in terms of milliseconds (msec).
Time Frame: Baseline, Day 4 (at 84 hrs)
Population: Safety population included all participants who began infusion with SAGE-547 injection.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
msec
  Change from Baseline at Day 4 (84 hrs):QT Interval | -28.5 (34.31)
  Change from Baseline at Day 4 (84 hrs):PR Interval | -1.0 (9.87)
  Change from Baseline at Day 4(84 hrs):QTc Interval | 13.3 (10.44)
  Change from Baseline at Day 4(84 hrs):QRS Duration | -3.5 (7.19)

19. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameter: Heart Rate
Description: ECGs parameter included heart rate expressed in terms of beats per minute (bpm).
Time Frame: Baseline, Day 4 (at 84 hrs)
Population: Safety population included all participants who began infusion with SAGE-547 injection.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
bpm | 14.3 (9.29)

20. Primary Outcome: Number of Participants With Physical Examination Findings
Description: Physical examinations included body weight, height, body mass index (BMI) and assessment of body systems (e.g., head, eyes, ears, nose, throat, lungs, abdomen, and extremities) as well as cognitive and mental health examinations (components of the neurological and psychiatric examinations, respectively).
Time Frame: At Day 4
Population: Safety population included all participants who began infusion with SAGE-547 injection.
Measure: Count of Participants; unit: Participants
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
Participants | 4

21. Primary Outcome: Number of Participants With Concomitant Medication Usage
Description: Concomitant medications are other prescription medications, over the counter (OTC) drugs or dietary supplements that a study participant takes in addition to the drug under investigation.
Time Frame: Baseline up to Day 11
Population: Safety population included all participants who began infusion with SAGE-547 injection.
Measure: Count of Participants; unit: Participants
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
Participants | 3

22. Primary Outcome: Number of Participants With Suicidal Ideation and Behavior as Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS scale consists of a baseline evaluation that assesses the lifetime experience of the participant with suicidal ideation and behavior, and a post-baseline evaluation that focuses on suicidality since the last study visit. The C-SSRS includes 'yes' or 'no' responses for assessment of suicidal ideation and behavior as well as numeric ratings for severity of ideation, (with score range from 1 to 5, higher score indicates more severity). The data was collected at time-points: Pre-infusion (Day 1 prior to dosing), Post-infusion (any time after the start of infusion on Day 1 up to 84 hrs).
Time Frame: Pre-infusion (Day 1 prior to dosing), Post-infusion (any time after the start of infusion on Day 1 up to 84 hrs)
Population: Efficacy population included all participants who began infusion with SAGE-547 injection and who completed at least 12 hours of infusion and have efficacy evaluations through the 12-hour visit.
Measure: Count of Participants; unit: Participants
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
Participants
  Pre-Infusion: Suicidal Ideation | 3
  Post-Infusion: Suicidal Ideation | 0
  Pre-Infusion: Suicidal Behavior | 1
  Post-Infusion: Suicidal Behavior | 0

23. Secondary Outcome: Maximum Plasma Concentration (Cmax) of SAGE-547
Time Frame: Predose (0 hrs), and 0.5, 1, 2, 3, 4, 6, 12, 24, 36, 40, 44, 48, 60, and 72 hrs post-dose
Population: Pharmacokinetic (PK) population included all who began infusion with SAGE-547 injection and for whom at least one evaluable PK sample was available.
Measure: Mean (Standard Deviation); unit: nanograms per millilter (ng/mL)
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
nanograms per millilter (ng/mL) | 97.2 (77.3)

24. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of SAGE-547
Description: Tmax is defined as the time at which Cmax of SAGE-547 occurred.
Time Frame: Predose (0 hrs), and 0.5, 1, 2, 3, 4, 6, 12, 24, 36, 40, 44, 48, 60, and 72 hrs post-dose
Population: PK population included all who began infusion with SAGE-547 injection and for whom at least one evaluable PK sample was available.
Measure: Median (Full Range); unit: hours
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
hours | 42 [12 to 48]

25. Secondary Outcome: Area Under the Concentration-Time Curve From Start of the Infusion Until the Time of the Last Sample (AUCall) of SAGE-547
Description: AUCall is defined as the area under the plasma SAGE-547 concentration time curves from the start of the infusion until the time the last sample was taken 72 hours later.
Time Frame: Predose (0 hrs), and 0.5, 1, 2, 3, 4, 6, 12, 24, 36, 40, 44, 48, 60, and 72 hrs post-dose
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: nanograms*hour per milliliter (ng*hr/mL)
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
nanograms*hour per milliliter (ng*hr/mL) | 3380 (1410)

26. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to 60 Hours (AUC0-60) of SAGE-547
Description: AUC0-60 is defined as the area under the plasma SAGE-547 concentration time curve during the intravenous infusion.
Time Frame: Predose (0 hrs), and 0.5, 1, 2, 3, 4, 6, 12, 24, 36, 40, 44, 48, and 60 hrs post-dose
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
ng*hr/mL | 3160 (1360)

27. Secondary Outcome: Area Under the Concentration-Time Curve in 24 Hours (AUC24) of SAGE-547
Description: AUC24 is defined as the area under the plasma SAGE-547 concentration-time curve in a 24-hour period during the maintenance dose.
Time Frame: Predose (0 hrs), and 0.5, 1, 2, 3, 4, 6, 12, and 24 hrs post-dose
Population: PK population included all who began infusion with SAGE-547 injection and for whom at least one evaluable PK sample was available. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | SAGE-547
Number analyzed (Participants) | 3
ng*hr/mL | 1590 (580)

28. Secondary Outcome: Average Drug Concentration in the Plasma at Steady State During a Dosing Interval (Cavg) of SAGE-547
Description: Cavg is defined as the plasma concentration of SAGE-547 at steady-state (average plasma concentration during the maintenance dose period; nominally 12 to 48 hrs).
Time Frame: From 12 to 48 hrs (36 hr of maintenance dose period)
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SAGE-547
Number analyzed (Participants) | 3
ng/mL | 66.1 (24.1)

29. Secondary Outcome: Plasma Clearance (CL) of SAGE-547
Description: Clearance of a drug was a measure of the rate at which a drug was metabolized or eliminated by normal biological processes.
Time Frame: Predose (0 hrs), and 0.5, 1, 2, 3, 4, 6, 12, 24, 36, 40, 44, 48, 60, and 72 hrs post-dose
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Liters per hour per kilogram (L/hr/kg)
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
Liters per hour per kilogram (L/hr/kg) | 1.08 (0.22)

30. Secondary Outcome: Change From Baseline in Hamilton Rating Scale for Depression-17 (HAM-D-17) Total Score
Description: The HAM-D-17 was used to rate the severity of depression in participants who were already diagnosed as depressed. The HAM-D-17 is comprised of 17 individual items: Items scored in a range of 0 to 2 include: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following items are scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis, where 0 indicated none/absent and higher scores indicated greater depression. The Total Score can range from 0 (least depression) to 52 (greater depression), and higher scores indicate a greater degree of depression. A negative change from baseline indicates less depression. A positive change from baseline indicates more depression.
Time Frame: Baseline, Day 1 (12 hrs), Day 2 (at 24 and 36 hrs), Day 3 (at 48 and 60 hrs), and Day 4 (at 84 hrs)
Population: Safety population included all participants who began infusion with SAGE-547 injection.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
score on a scale
  Change From Baseline at Day 1 (12 hrs) | -21.8 (5.50)
  Change From Baseline at Day 2 (24 hrs) | -23.3 (4.19)
  Change From Baseline at Day 2 (36 hrs) | -24.8 (3.59)
  Change From Baseline at Day 3 (48 hrs) | -24.3 (4.99)
  Change From Baseline at Day 3 (60 hrs) | -24.8 (4.19)
  Change From Baseline at Day 4 (84 hrs) | -21.3 (6.85)

31. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I) Score
Description: The CGI-I response was defined as having a score of 1 (very much improved) or 2 (much improved). CGI-I assessment employs a 7-point Likert scale to measure the improvement in the participant's condition. The investigator rated the participant's total improvement whether or not it was due entirely to drug treatment. Response choices include: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. The CGI-I was only rated at post-treatment assessments. By definition, all CGI-I assessments were evaluated against baseline conditions.
Time Frame: Day 1 (12 hrs), Day 2 (at 24 and 36 hrs), on Day 3 (at 48 and 60 hrs), and Day 4 (at 84 hrs)
Population: Efficacy population included all participants who began infusion with SAGE-547 injection and who completed at least 12 hours of infusion and had efficacy evaluations through the 12-hour visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAGE-547
Number analyzed (Participants) | 4
score on a scale
  Day 1 (12 hrs) | 1.8 (0.50)
  Day 2 (24 hrs) | 1.3 (0.50)
  Day 2 (36 hrs) | 1.0 (0.00)
  Day 3 (48 hrs) | 1.3 (0.50)
  Day 3 (60 hrs) | 1.3 (0.50)
  Day 4 (84 hrs) | 1.5 (0.58)

ADVERSE EVENTS:
Time Frame: AEs: Up to Day 11; SAEs: Up to Day 34
Description: Safety population included all participants who began infusion with SAGE-547 injection.
Groups:
- SAGE-547: Participants received SAGE-547 intravenous injection over 60 hours (including 12-hour titration infusion of 21.5 micrograms/kg/hr [4 hrs], 43 micrograms/kg/hr [4 hrs] and 64.5 micrograms/kg/hr [4 hrs] on Day 1, followed by 13 to 48 hrs [36 hrs] maintenance infusion of 86 micrograms/kg/hr from Day 1 to 3, followed by a 12-hr taper infusion of 64.5 micrograms/kg/hr [49 - 52 hrs], 43 micrograms/kg/hr [53 - 56 hrs] and 21.5 micrograms/kg/hr [57 - 60 hrs] on Day 3).
Arm/Group | SAGE-547
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SAGE-547 (N=4)
Infusion Site Discomfort (General disorders) | 1
Infusion Site Erythema (General disorders) | 1
Infusion Site Pain (General disorders) | 1
Blood Thyroid Stimulating Hormone Increased (Investigations) | 1
Dizziness (Nervous system disorders) | 1
Sedation (Nervous system disorders) | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can either be a party and subject to the same restrictions as the institution, or if not a party, the restrictions are described on the face of the contract (i.e., PI is a contractor of the institution; PI is part of a larger group of study personnel; institution has contracted with or otherwise bound all study personnel under confidentiality obligations and requirements to vest intellectual property to the institution).